CLINICAL TRIAL: NCT03133481
Title: Adductor Canal Block Versus Femoral Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Promil Kukreja, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F140917004
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Arthropathy of Knee
Keywords: Adductor Canal Block; Femoral Canal Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The first two groups will have 50 participants each (100 total) the "Adductor Canal Nerve Catheter" group and the "Femoral Nerve Catheter," group. Participants will be randomized using block randomization. The blocks will be assigned randomly based on computer generated numbers.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Adductor Canal Nerve Block (Active Comparator): Participants will be randomized using block randomization.
  Interventions: Procedure: Adductor Canal Nerve Block
- Femoral Nerve Block (Active Comparator): Participants will be randomized using block randomization.
  Interventions: Drug: Femoral Nerve Block

INTERVENTIONS:
Procedure: Adductor Canal Nerve Block — Adductor Canal never technique
  Other Names: ropivacaine
  Arms: Adductor Canal Nerve Block
Drug: Femoral Nerve Block — Traditional technique
  Other Names: ropivacaine
  Arms: Femoral Nerve Block

SUMMARY:
Peripheral nerve blocks catheters of the femoral nerve have long been used for perioperative analgesia in total knee arthroplasty (TKA). These blocks provide effective analgesia and patient satisfaction for surgical pain relief. However, one of the main drawbacks to the femoral nerve block (FNB) is a denser motor block of the quadriceps muscle that can delay aggressive physical therapy and subsequent recovery from surgery. (1) Recently, there has been increasing interest in performing adductor canal blocks (ACB) with the aim of less motor blockade while providing commensurate analgesia compared to the FNB. (1,2) Current investigative reports have provided only preliminary data, and there is potential to change the standard of care for TKA as more data mounts in favor of ACBs. The goal of this study is to verify the analgesic equivalence of the two blocks, compare patient satisfaction, surgeon satisfaction, and physical therapy grading between the two blocks. Potentially, this would change the standard of care for TKA patients at this institution.

DETAILED DESCRIPTION:
The specific objectives of this study are to determine the effectiveness of ACB for analgesia compared to FNB as determined by patient reported VAS scores. Determine the effectiveness of ACB for analgesia compared to FNB as determined by opioid usage. Determine the effectiveness of ACB in physical therapy as determined by early ambulation distance. Determine the surgeon satisfaction via survey, and determine if there is any difference in time to discharge between the two blocks.

Participants in the investigational group will received an adductor canal nerve catheter prior to TKA surgery. Participants in the control group will receive a femoral nerve catheter prior to TKA surgery. After surgery, the patient will be seen in the recovery room to bolus the catheters and start continuous infusions of ropivacaine.

The primary endpoints include, Pain Scores (VAS) at immediate post op, 24 hours, and 48 hours, including highest, opioid consumption at 24 hours and 48 hours pain score at any given time post operatively, physical therapist assessment of patient participation 0-100, distance ambulated at 24 to 48 hours, patient satisfaction, surgeon satisfaction, and hours to discharge.

Participants will be recruited, identified, and interviewed by either the study Principal Investigator or one of the co-investigators. The interviewing investigator will confirm eligibility and the absence of any exclusionary criteria. Details of the study (including risks) will be explained to prospective participants to their satisfaction and consent forms will then be signed.

Randomization: Upon enrollment into the study, participants will be randomized 1:1 to either the investigational group (adductor canal nerve catheter) or the control group (femoral nerve catheter). Randomization will be performed using a random number generator Participants in this study will be randomized into two interventional groups. The participant in the "adductor canal nerve catheter" investigational group will receive an adductor canal block catheter placed under direct ultrasound guidance. The participants in the "femoral nerve catheter" control group will receive a femoral nerve clock catheter placed under direct ultrasound guidance with a stimulating needle. Investigational group participants in the adductor canal block arm will receive an adductor canal block catheter placed under direct ultrasound guidance as follows. Patients will be placed supine with their block limb supinated about 20 degrees to facilitate access to the anteromedial thigh. Standard noninvasive monitors will be applied, and oxygen administered via nasal canula. Parenteral midazolam and fentanyl will be titrated to patient comfort.

Standard skin sterilization, prepping, and draping will be applied to the area. Under ultrasound guidance the needle will be advanced into the adductor canal. After negative aspiration, a bolus of 20 ml 0.5% Ropivacaine will be injected under direct visualization in 5 mL aliquots ensuring proper placement of the needle tip. The catheter will be advanced in this position at least 2 cm and not more than 5 cm and secured to the skin with tegaderm. Patients will be evaluated immediately post-operatively in the PACU (Post anesthesia care unit) to determine VAS score from 0-10.

Patients will be given a standard pain regimen while in the hospital. 24 hour opioid consumption will be calculated. Patients will be evaluated 24 and 48 hours post operatively for VAS score, duration of sensory and motor block, and patient satisfaction from 0-10. The catheter will be removed on post operative day 2. Patient will be followed up until nerve block resolved. Physical therapists in the hospital will be surveyed with a standard questionnaire regarding the patients ability to participate in physical therapy sessions on a scale of 0-10. Ambulation distance at 24 and 48 hours will be recorded per their notes. The surgeons performing the procedures will be surveyed in a general sense regarding their impression of patient recovery with this block. The hours to discharge will be calculated.

Control group participants in the femoral nerve block arm will receive a femoral nerve block catheter placed under direct ultrasound guidance with the stimulating needle as follows. Patients will be placed supine with their block limb exposed to facilitate access to the anterior inguinal area. Standard noninvasive monitors will be applied, and oxygen administered via nasal canula. Parenteral midazolam and fentanyl will be titrated to patient comfort. Standard skin sterilization, prepping, and draping will be applied to the area. Under ultrasound guidance the needle will be advanced to the femoral nerve. After negative aspiration, a bolus of 20 ml 0.5% Ropivacaine will be injected under direct visualization in 5 mL aliquots ensuring proper placement of the needle tip. The catheter will be advanced in this position at least 2 cm and not more than 5 cm and secured to the skin with tegaderm. Patients will be evaluated immediately post-operatively in the PACU (Post anesthesia care unit) to determine VAS score from 0-10.

Physical therapist and physicians will be asked to complete a short survey after their patient has enrolled in the study. A Waiver of Informed Consent is requested for their participation.

Patients will be given a standard pain regimen while in the hospital. 24 hour opioid consumption will be calculated. Patients will be evaluated 24 and 48 hours post operatively for VAS score, duration of sensory and motor block, and patient satisfaction from 0-10. The catheter will be removed on post operative day 2. Patient will be followed up until nerve block resolved. Physical therapists in the hospital will be surveyed with a standard questionnaire regarding the patients ability to participate in physical therapy sessions on a scale of 0-100. Ambulation distance at 24 and 48 hours will be recorded per their notes. The surgeons performing the procedures will be surveyed in a general sense regarding their impression of patient recovery with this block then the hours will be calculated to the hours to discharge for each patient.

All demographic and clinical variables with continuous measures will be expressed as means and standard deviations; categorical factors will be expressed as proportions. For non-normal data, the medians and inter quartile ranges will be displayed. The distribution of the continuous factors will be examined using the Kolmogorov-Smirnov test. For data that are normally distributed, the one-way ANOVA and Student's t-test will be used to compare groups of data. For data that are not normally distributed, the Kruskal-Wallis and Mann-Whitney tests will be used for comparisons. Chi-square and Fisher's exact tests will be used to analyze categorical data. For all comparisons, a value of p < 0.05 will be considered statistically significant.

Primary Outcome Analysis: Statistical analyses will be performed using SAS for Windows, version 9.2. Student's t-test will be used to compare post-operative pain scores for investigational and control subjects. Linear regression will be also be used to test the relationship between pain scores and regional anesthetic technique, while controlling for relevant clinical and demographic variables. Distance of first ambulation will be analyzed using Cox proportional hazards model. Student's t-test will be used to compare patient and surgeon satisfaction.

Statistical Power and Sample Size Estimates: Sample size (94) was determined using a Cohen's d table assuming a mean pain VAS score of 8 (sd = 3) on a scale of 0-10 for control subjects. A sample of 94 participants (45 patients in the adductor canal block group, and 49 patients in the femoral nerve block group) will have approximately 80% power to detect a reduction in pain score of at least 50%, and approximately 99% to detect an 80% reduction in pain score.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing total knee arthroplasty with regional anesthesia planned for postoperative analgesia.
* Adult, 19 years of age or older
* Patient classified as American Society of Anesthesiology (ASA) class I, II, or III

Exclusion Criteria:

* Any subject not classified as an ASA I, II, or III
* Allergy/intolerance to local anesthetic
* Pre-existing neurologic or anatomic deficit in lower extremity on the side of the surgical site
* Coexisting coagulopathy such as hemophilia or von Willebrand disease

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Promil Kukreja, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Started | 45 | 49
Completed | 45 | 45
Not Completed | 0 | 4
Not completed — FC Catheter fell out post operative day1 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block | Total
Number analyzed (Participants) | 45 | 49 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 21 | 49
  >=65 years | 17 | 28 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.01) | 65.4 (9.28) | 64.4 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45 | 49 | 94

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance Ambulated at 24 Hours Post Operatively
Description: Distance ambulated in feet from the end of surgery to 24 hours postoperatively
Time Frame: Baseline up to 24 hours after the Anesthesia Record Stop Time
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
feet | 70.2 (66.94) | 48.44 (45.76)

2. Primary Outcome: Mean Distance Ambulated at 48 Hours Post Operatively
Description: Distance ambulated in feet from the end of surgery to 48 hours postoperatively
Time Frame: From the Anesthesia Record Stop Time to 48 hours after the Anesthesia Record Stop Time
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
feet | 129.02 (92.33) | 106.38 (83.39)

3. Secondary Outcome: Mean Pain Scores Immediately Preoperatively
Description: Visual Analog Scale (VAS) score immediately preoperatively.
  The Visual Analog Scale is a standard numerical pain score reported by the patient, from 0-10, where 0=no pain, and 10=worst pain.
Time Frame: baseline up to time of anesthesia record start time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
score on a scale | 3.07 (3.43) | 3.38 (3.44)

4. Secondary Outcome: Mean Opioid Consumption as Measured by Oral Morphine Milligram Equivalents
Description: Preoperatively, opioid consumption will be measured from baseline to the Anesthesia Record Start Time in Oral Morphine Equivalents
Time Frame: from baseline to two hours
Measure: Mean (Standard Deviation); unit: Oral Morphine Milligram Equivalents
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
Oral Morphine Milligram Equivalents | 23 (8.52) | 22.33 (8.23)

5. Secondary Outcome: Patient Satisfaction at 48 Hours Post Operatively
Description: Patient satisfaction score, on an analog scale from 0-10, with 0 being the lowest satisfaction and 10 being the highest satisfaction.
Time Frame: Baseline up to 48 hrs
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
score on a scale | 8.71 (2.16) | 9.24 (1.26)

6. Secondary Outcome: Mean Hours to Discharge
Description: Mean hours to discharge, from the time of admittance to the time of discharge
Time Frame: Baseline to discharge (approximately 90 hrs)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
hours | 89.66 (32.24) | 83.78 (14.52)

7. Secondary Outcome: Mean Pain Scores in PACU
Description: The Mean Pain Score (VAS) at no more than 4 hours after the Anesthesia Record Stop Time.
  The Visual Analog Scale is a standard numerical pain score reported by the patient, from 0-10, where 0=no pain, and 10=worst pain.
Time Frame: Immediately post operatively, not more than 4 hours after pacu admittance
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
score on a scale | 3.91 (3.19) | 2.98 (3.05)

8. Secondary Outcome: Mean Pain Scores at 24 Hours
Description: Visual Analog Scale (VAS) score at 24 hours from the time of Anesthesia Record Stop Time.
  The Visual Analog Scale is a standard numerical pain score reported by the patient, from 0-10, where 0=no pain, and 10=worst pain.
Time Frame: From the Anesthesia Record stop time to 24 hours after Anesthesia Record stop time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
score on a scale | 4.18 (2.64) | 4 (2.35)

9. Secondary Outcome: Mean Pain Scores 48 Hours Postoperatively
Description: Visual Analog Scale (VAS) score at 48 hours from the time of Anesthesia Record Stop Time.
  The Visual Analog Scale is a standard numerical pain score reported by the patient, from 0-10, where 0=no pain, and 10=worst pain.
Time Frame: From the Anesthesia Record Stop Time to 48 hours from the Anesthesia Record Stop Time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
score on a scale | 4.53 (2.37) | 4.44 (2.29)

10. Secondary Outcome: Mean Opioid Consumption as Measured in Oral Morphine Milligram Equivalents
Description: Mean opioid consumption as measured immediately post operatively from Anesthesia Record Stop Time to 4 hours after Anesthesia Record Stop Time in Oral Morphine Milligram Equivalents
Time Frame: Post operatively through 4 hours
Measure: Mean (Standard Deviation); unit: Oral Morphine Milligram Equivalents
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
Oral Morphine Milligram Equivalents | 53.92 (34.56) | 50.77 (32.99)

11. Secondary Outcome: Mean Opioid Consumption as Measured in Oral Morphine Milligram Equivalents
Description: Mean opioid consumption as calculated from the time of Anesthesia Record Stop Time to 24 hours after Anesthesia Record Stop Time in Oral Morphine Equivalents
Time Frame: From immediately post operatively through 24 hours
Measure: Mean (Standard Deviation); unit: Oral Morphine Milligram Equivalents
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
Oral Morphine Milligram Equivalents | 75.54 (49.81) | 68.78 (55.08)

12. Secondary Outcome: Mean Opioid Consumption as Measured in Oral Morphine Equivalents
Description: Mean opioid consumption as calculated from Anesthesia Record Stop Time to 48 hours after Anesthesia Record Stop Time in Oral Morphine Milligram Equivalents
Time Frame: From immediately post operatively through 48 hours
Measure: Mean (Standard Deviation); unit: Oral Morphine Milligram Equivalents
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
Number analyzed (Participants) | 45 | 45
Oral Morphine Milligram Equivalents | 55.49 (32.3) | 44.47 (22.26)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Adductor Canal Nerve Block | Femoral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/49
Other Adverse Events (participants affected / at risk) | 0/45 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03133481/Prot_SAP_000.pdf